CLINICAL TRIAL: NCT07192601
Title: Developing an E-Cigarette Cessation Intervention for Hispanic/Latina(o) Youth in Florida
Brief Title: Developing an E-Cigarette Cessation Intervention for Hispanic/Latina(o) Youth in Florida: The BReATHE Study
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Florida International University (Other)
Collaborators: James and Esther King Biomedical Research Program (Other)
Responsible Party: Principal Investigator, Elisa M. Trucco, PhD, Associate Professor of Psychology, Florida International University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB-24-0113; 24K09 (Other Grant/Funding Number: Florida Department of Health)
Record Dates: First submitted 2025-09-05; First posted 2025-09-25 (Actual); Last update posted 2025-09-25 (Actual); Status verified 2025-09

CONDITIONS: Vaping Teens; Vaping Behaviors; Vaping Cessation; Tobacco Use Disorder
Keywords: adolescents; vaping cessation; cognitive behavioral therapy
MeSH Terms: conditions — Tobacco Use Disorder

STUDY DESIGN:
Intervention Model Description: As this is a pilot study, all participants (N=120) will be enrolled in the same vaping cessation program, which will be grounded in an empirically supported psychosocial smoking cessation program (i.e., Cognitive Behavioral Therapy, CBT) that has been found to be effective in both adults, as well as adolescents.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single Arm (Other): See Intervention Section
  Interventions: Behavioral: E-cigarette Cessation Manual

INTERVENTIONS:
Behavioral: E-cigarette Cessation Manual — E-cigarette cessation manual development. Empirically supported treatment content. We anticipate grounding the intervention in an empirically supported psychosocial smoking cessation program (i.e., Cognitive Behavior Therapy; CBT), which has been found to be effective with both adults and adolescents to quit cigarette smoking (Vinci, 2020). We anticipate including sessions that teach CBT skills to help adolescents quit e-cigarette use. These CBT skills and format will be adapted from prior manualized CBT smoking cessation interventions for adolescent smoking cessation and manualized CBT e-cigarette intervention for adolescents and young adults that are currently ongoing (e.g., Kong et al., 2017; Kong et al., 2021; Bold et al., 2022). The structure and content of the e-cigarette cessation manual will be further informed by themes and sub-themes from the focus group data analysis relating to both surface and deep structure cultural modifications.

SUMMARY:
Investigators will create and implement an e-cigarette intervention for Hispanic/Latino (H/L) high school youth. Focus groups with the target population (i.e., H/L high school students) and meetings with a community advisory board (CAB) will inform this intervention. The intervention will be tested with 120 H/L high school e-cigarette users to assess feasibility and promise for reducing use.

DETAILED DESCRIPTION:
The e-cigarette cessation intervention will be grounded in an empirically supported psychosocial smoking cessation program (i.e., Cognitive Behavioral Therapy, CBT; Cavallo et al., 2007; Krishnan-Sarin et al., 2013; Vinci et al., 2020) that has been found to be effective in both adults, as well as adolescents. The CBT intervention will likely include a total of 6 weekly sessions adapted for e-cigarettes that will be developed by the investigators and in consultation with a community advisory board. Based on initial feedback from focus groups, the sessions will likely take place in person, be in a group format, and be no longer than 50 minutes in duration. Some sessions will also include the adolescents' caregivers. We propose a "Preparation to Quit" session conducted approximately one week prior to quitting, which incorporates motivational strategies and assistance to aid quitting, set a quit day, and make a quit plan. This will be followed by a "pre-quit" session on the day before the quit day to review the quit plan, and then an additional session after the quit day that will focus on: 1) coping with cravings and withdrawal symptoms and identifying high risk situations, 2) becoming assertive, developing refusal skills, 3) stress/anger management skills, 4) problem-solving skills, 5) enhancing communication and family dynamics, 6) behavioral activation and community reinforcement, and 7) relapse prevention and coping with lapses. Session content and format will be adapted to be culturally relevant and integrate needs and strengths that are gleaned from focus groups. In addition to attending sessions, participants will be asked to complete an in-person baseline questionnaire session (~1hr) and a salivary cotinine assessment to objectively quantify recent nicotine exposure to verify current e-cigarette usage prior to their first cessation session. Participants will also be asked to complete a weekly 5-minute online survey on REDCap reflecting past week substance use. Participants will complete a salivary cotinine assessment to objectively quantify nicotine exposure during their last intervention session. Participants will also be asked to complete a follow-up questionnaire session (30 minutes) three months after they have completed the intervention, as well as a salivary cotinine assessment.

ELIGIBILITY:
Inclusion Criteria:

* Enrolled in high school or 14-18 years old
* Identify as being of Hispanic/Latino origin
* Report past month e-cigarette use and verified by saliva cotinine test

Exclusion Criteria:

* having a history of severe psychiatric conditions (e.g., bipolar disorder)
* currently enrolled in or planning on enrolling in another e-cigarette and/or tobacco cessation intervention
* having potential difficulties comprehending study procedures (e.g., not able to speak/write in English or Spanish, have a severe learning disability)

Ages: 14 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 120 (Estimated)
Dates: Start 2024-05-01 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2028-04-30 (Estimated)

PRIMARY OUTCOMES:
E-Cigarette Assessment for Youth-Revised checklist | Baseline assessment: data will be reported on past 1-month and 1-year e-cigarette use Each weekly intervention session: data will be reported on past 1-week e-cigarette use Follow-up assessment: data will be reported on past 1-month e-cigarette use
  This measure assesses the timing, brand, flavoring, quantity, and frequency of current and past e-cigarette use.
Salivary cotinine samples | Saliva cotinine samples that can detect past-week nicotine use will be obtained at Baseline (Week 0), at the end of treatment (Week 6), and at the 3-month follow-up after treatment completion (Week 18).
  To biochemically verify self-reports of abstinence, saliva samples will be obtained using NicAlert cotinine test strips.
Patient-Reported Outcomes Measurement Information System Nicotine Dependence Bank for E-Cigarettes | Baseline assessment: data will be reported on past 1-month symptoms Each weekly intervention session: data will be reported on past 1-week symptoms Follow-up assessment: data will be reported on past 1-month symptoms
  The Patient-Reported Outcomes Measurement Information System Nicotine Dependence Bank for E-Cigarettes (PROMIS-E) is a 4-item measure (each item scored on a 5-point Likert scale) that assesses nicotine dependence. Values range from 0 to 16 with higher scores representing worse outcomes.
Questionnaire of Vaping Craving | Baseline assessment: data will be reported on past 1-month craving Each weekly intervention session: data will be reported on past 1-week craving Follow-up assessment: data will be reported on past 1-month craving
  The Questionnaire of Vaping Craving (QVC) is a 10-item measure (each item scored on a 7-point Likert scale) that assesses vaping craving. Values range from 10 to 70 with higher scores representing worse outcomes.
Wisconsin Smoking Nicotine Withdrawal Scale | Baseline assessment: data will be reported on past 1-week withdrawal symptoms Each weekly intervention session: data will be reported on past 1-week withdrawal symptoms Follow-up assessment: data will be reported on past 1-week withdrawal symptoms
  The Wisconsin Smoking Nicotine Withdrawal Scale (WSWS) is a 28-item measure (each item scored on a 5-point Likert scale) that assesses nicotine withdrawal symptoms. Values range from 0 to 112 with higher scores representing worse outcomes.

SECONDARY OUTCOMES:
Timeline Followback questionnaire | Baseline assessment: data will be reported on past 1-month and past 1-year substance use Each weekly intervention session: data will be reported on past 1-week substance use Follow-up assessment: data will be reported on past 1-month substance use
  Frequency and quantity of current and past use of other substances beyond e-cigarettes (e.g., other tobacco products, alcohol, cannabis) will also be queried.
Adolescent E-Cigarette Consequences Questionnaire | Baseline assessment: data will be reported on past 1-week expectancies Follow-up assessment: data will be reported on past 1-week expectancies
  The Adolescent E-Cigarette Consequences Questionnaire (AECQ) is a 31-item measure (each item scored on a 5-point Likert scale) that assesses outcome expectancies when using an e-cigarette. Values range from 31 to 155 with higher scores representing worse outcomes.
PROMIS Emotional Distress Depression and Anxiety Pediatric Item Bank | Baseline assessment: data will be reported on past 2-week symptoms experienced Follow-up assessment: data will be reported on past 2-week symptoms experienced
  This is a 5-item measure (each item scored on a 5-point Likert scale) that assesses symptoms of depression and anxiety. Values range from 0 to 20 with higher scores representing worse outcomes.
Parental Monitoring, Child Disclosure, and Relationship Quality | Baseline assessment: data will be reported on past 1-week perceptions Follow-up assessment: data will be reported on past 1-week perceptions
  This 22-item measure (each item scored on a 5-point Likert scale) assesses parental monitoring, child disclosure, and relationship quality. Values range from 0 to 88 with higher scores representing better outcomes.
Resistance to Peer Influence | Baseline assessment: data will be reported on past 1-week perceptions Follow-up assessment: data will be reported on past 1-week perceptions
  The Resistance to Peer Influence (RPI) is a 10-item measure (each item scored on a 4-point Likert scale) that assesses an adolescent's ability to resist peer influence across multiple hypothetical scenarios. Values range from 0 to 40 with higher scores representing better outcomes.
Multidimensional Scale of Perceived Social Support | Baseline assessment: data will be reported on past 1-week perceptions Follow-up assessment: data will be reported on past 1-week perceptions
  Social support (e.g., friends, family members) will be measured by this 12-item (each item scored on a 7-point Likert scale) measure. Values range from 12 to 84 with higher scores representing better outcomes.
Treatment Acceptability | Final weekly intervention session: data will be reported on past 2-month general impressions with the treatment.
  Participants will complete a survey encompassing multiple-choice questions and open-ended text boxes regarding their satisfaction with the vaping cessation program.

CONTACTS AND LOCATIONS:
Locations (1):
- FIU Center for Children and Families, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: Undecided
To enhance the value and further the advancement of this research, we will consider sharing information collected from participants with other qualified individuals within the scientific community on a case-by-base basis while safeguarding the confidentiality/privacy of participants. Our underlying philosophy is to widely distribute, disseminate, and share all derived data and resources.

REFERENCES:
- [Background] Bastiaens L, Galus J. The DSM-5 Self-Rated Level 1 Cross-Cutting Symptom Measure as a Screening Tool. Psychiatr Q. 2018 Mar;89(1):111-115. doi: 10.1007/s11126-017-9518-7. PMID 28523431
- [Background] Benowitz NL, Bernert JT, Caraballo RS, Holiday DB, Wang J. Optimal serum cotinine levels for distinguishing cigarette smokers and nonsmokers within different racial/ethnic groups in the United States between 1999 and 2004. Am J Epidemiol. 2009 Jan 15;169(2):236-48. doi: 10.1093/aje/kwn301. Epub 2008 Nov 19. PMID 19019851
- [Background] Bold K, Kong G, Cavallo D, Davis D, Jackson A, Krishnan-Sarin S. School-based E-cigarette cessation programs: What do youth want? Addict Behav. 2022 Feb;125:107167. doi: 10.1016/j.addbeh.2021.107167. Epub 2021 Oct 28. PMID 34753093
- [Background] Cavallo DA, Cooney JL, Duhig AM, Smith AE, Liss TB, McFetridge AK, Babuscio T, Nich C, Carroll KM, Rounsaville BJ, Krishnan-Sarin S. Combining cognitive behavioral therapy with contingency management for smoking cessation in adolescent smokers: a preliminary comparison of two different CBT formats. Am J Addict. 2007 Nov-Dec;16(6):468-74. doi: 10.1080/10550490701641173. PMID 18058412
- [Background] Cristello JV, Sutherland MT, Trucco EM. A preliminary validation of the adolescent e-cigarette consequences questionnaire. Drug Alcohol Depend. 2020 Aug 1;213:108118. doi: 10.1016/j.drugalcdep.2020.108118. Epub 2020 Jun 12. PMID 32559666
- [Background] Dowd AN, Motschman CA, Tiffany ST. Development and Validation of the Questionnaire of Vaping Craving. Nicotine Tob Res. 2019 Jan 1;21(1):63-70. doi: 10.1093/ntr/nty046. PMID 29546379
- [Background] Hartmann SA, Cristello JV, Manresa O, Trucco EM. The e-cigarette assessment for youth-Revised (EAsY-R): Preliminary results of a pilot study of measure refinement via cognitive interviewing. J Res Adolesc. 2024 Sep;34(3):845-856. doi: 10.1111/jora.12957. Epub 2024 Apr 28. PMID 38679807
- [Background] Hughes JR, Keely JP, Niaura RS, Ossip-Klein DJ, Richmond RL, Swan GE. Measures of abstinence in clinical trials: issues and recommendations. Nicotine Tob Res. 2003 Feb;5(1):13-25. PMID 12745503
- [Background] Kong G, Bold KW, Cavallo DA, Davis DR, Jackson A, Krishnan-Sarin S. Informing the development of adolescent e-cigarette cessation interventions: A qualitative study. Addict Behav. 2021 Mar;114:106720. doi: 10.1016/j.addbeh.2020.106720. Epub 2020 Oct 21. PMID 33162230
- [Background] Kong G, Goldberg AL, Dallery J, Krishnan-Sarin S. An open-label pilot study of an intervention using mobile phones to deliver contingency management of tobacco abstinence to high school students. Exp Clin Psychopharmacol. 2017 Oct;25(5):333-337. doi: 10.1037/pha0000151. PMID 29048181
- [Background] Krishnan-Sarin S, Cavallo DA, Cooney JL, Schepis TS, Kong G, Liss TB, Liss AK, McMahon TJ, Nich C, Babuscio T, Rounsaville BJ, Carroll KM. An exploratory randomized controlled trial of a novel high-school-based smoking cessation intervention for adolescent smokers using abstinence-contingent incentives and cognitive behavioral therapy. Drug Alcohol Depend. 2013 Sep 1;132(1-2):346-51. doi: 10.1016/j.drugalcdep.2013.03.002. Epub 2013 Mar 22. PMID 23523130
- [Background] Morean ME, Krishnan-Sarin S, S O'Malley S. Assessing nicotine dependence in adolescent E-cigarette users: The 4-item Patient-Reported Outcomes Measurement Information System (PROMIS) Nicotine Dependence Item Bank for electronic cigarettes. Drug Alcohol Depend. 2018 Jul 1;188:60-63. doi: 10.1016/j.drugalcdep.2018.03.029. Epub 2018 Apr 26. PMID 29753155
- [Background] Sobell LC, Cunningham JA, Sobell MB. Recovery from alcohol problems with and without treatment: prevalence in two population surveys. Am J Public Health. 1996 Jul;86(7):966-72. doi: 10.2105/ajph.86.7.966. PMID 8669520
- [Background] Stattin H, Kerr M. Parental monitoring: a reinterpretation. Child Dev. 2000 Jul-Aug;71(4):1072-85. doi: 10.1111/1467-8624.00210. PMID 11016567
- [Background] Steinberg L, Monahan KC. Age differences in resistance to peer influence. Dev Psychol. 2007 Nov;43(6):1531-1543. doi: 10.1037/0012-1649.43.6.1531. PMID 18020830
- [Background] Vinci C. Cognitive Behavioral and Mindfulness-Based Interventions for Smoking Cessation: a Review of the Recent Literature. Curr Oncol Rep. 2020 May 16;22(6):58. doi: 10.1007/s11912-020-00915-w. PMID 32415381
- [Background] Welsch SK, Smith SS, Wetter DW, Jorenby DE, Fiore MC, Baker TB. Development and validation of the Wisconsin Smoking Withdrawal Scale. Exp Clin Psychopharmacol. 1999 Nov;7(4):354-61. doi: 10.1037//1064-1297.7.4.354. PMID 10609970
- [Background] Zimet GD, Powell SS, Farley GK, Werkman S, Berkoff KA. Psychometric characteristics of the Multidimensional Scale of Perceived Social Support. J Pers Assess. 1990 Winter;55(3-4):610-7. doi: 10.1080/00223891.1990.9674095. PMID 2280326